CLINICAL TRIAL: NCT00344903
Title: Longitudinal Cohort Study of Dallas County Residents to Identify Novel Determinants of Atherosclerotic Heart Disease: The DHS 2
Brief Title: Dallas Heart Study 2: Return Clinic Visit for the Dallas Heart Study Cohort
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Donald W. Reynolds Foundation (Other)
Responsible Party: Helen Hobbs, MD, UT Southwestern Medical Center
Other Study IDs: DHS-2-001
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2009-02

CONDITIONS: Atherosclerosis; Congestive Heart Failure; Left Ventricular Hypertrophy; Diabetes Mellitus; Hypertension; Obesity; Metabolic Syndrome X; Myocardial Infarction
Keywords: Atherosclerosis; Heart Failure; Ventricular Hypertrophy; Myocardial Infarction; Screening; Hypertension; Diabetes; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Atherosclerosis; Heart Failure; Hypertrophy, Left Ventricular; Diabetes Mellitus; Hypertension; Obesity; Metabolic Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Serum DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Dallas Heart Study (DHS-1) is a large, multi-ethnic, population-based epidemiological study designed to identify determinants of atherosclerotic heart disease (ASHD) in a representative United States (US) urban environment. This study completed enrollment in 2003.

Our objective is to pinpoint factors contributing to progression:

1. from health to ASHD risk;
2. from ASHD risk to subclinical ASHD; and
3. from subclinical to clinical ASHD.

Identification of the critical factors in these transitions will enable targeted implementation of appropriate therapy to interdict before clinical ASHD develops.

DETAILED DESCRIPTION:
Early medical intervention in asymptomatic individuals at risk is the most effective strategy to combat atherosclerotic heart disease (ASHD). The major roadblock to effective ASHD prevention is that conventional tools to assess ASHD risk are inadequate and new methods are needed to identify susceptible individuals before the disease process is established. Other successful public-health screening programs have incorporated direct imaging procedures (e.g. mammography, colonoscopy); yet in ASHD, direct imaging of the vasculature has not been incorporated into the risk stratification algorithms.

The Dallas Heart Study (DHS-1) is a large, multi-ethnic, population-based epidemiological study designed to identify determinants of ASHD in a representative US urban environment. This study completed enrollment in 2003.

In DHS-2 we will transform the Dallas Heart Study from a cross-sectional health survey (DHS-1) into a longitudinal cohort study (DHS-2). We will perform state-of-the-art cardiovascular (CV) imaging coupled to biomarkers, genetic markers and classical ASHD risk factors. We will repeat the detailed clinical phenotyping performed between 2000-2003 to capture interval changes in ASHD risk and disease burden. Our objective is to pinpoint factors contributing to progression:

1. from health to ASHD risk;
2. from ASHD risk to subclinical ASHD; and
3. from subclinical to clinical ASHD.

Identification of the critical factors in these transitions will enable targeted implementation of appropriate therapy to interdict before clinical ASHD develops.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-70
* Participant in DHS-1 study completing visit 2 (blood sampling) and visit 3 (clinic visit)
* Provision of informed consent

Exclusion Criteria:

* None--population study

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who participated in DHS-1. The study will include equal numbers of men and women and will include 50% African Americans
Sampling Method: Probability Sample
Enrollment: 3400 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Hobbs, MD, Study Chair — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Victor RG, Haley RW, Willett DL, Peshock RM, Vaeth PC, Leonard D, Basit M, Cooper RS, Iannacchione VG, Visscher WA, Staab JM, Hobbs HH; Dallas Heart Study Investigators. The Dallas Heart Study: a population-based probability sample for the multidisciplinary study of ethnic differences in cardiovascular health. Am J Cardiol. 2004 Jun 15;93(12):1473-80. doi: 10.1016/j.amjcard.2004.02.058. PMID 15194016
- [Derived] Kay FU, Abbara S, Joshi PH, Garg S, Khera A, Peshock RM. Identification of High-Risk Left Ventricular Hypertrophy on Calcium Scoring Cardiac Computed Tomography Scans: Validation in the DHS. Circ Cardiovasc Imaging. 2020 Feb;13(2):e009678. doi: 10.1161/CIRCIMAGING.119.009678. Epub 2020 Feb 18. PMID 32066275
- [Derived] Rader F, Franklin SS, Mirocha J, Vongpatanasin W, Haley RW, Victor RG. Superiority of Out-of-Office Blood Pressure for Predicting Hypertensive Heart Disease in Non-Hispanic Black Adults. Hypertension. 2019 Nov;74(5):1192-1199. doi: 10.1161/HYPERTENSIONAHA.119.13542. Epub 2019 Sep 16. PMID 31522619
- [Derived] Garg S, de Lemos JA, Matulevicius SA, Ayers C, Pandey A, Neeland IJ, Berry JD, McColl R, Maroules C, Peshock RM, Drazner MH. Association of Concentric Left Ventricular Hypertrophy With Subsequent Change in Left Ventricular End-Diastolic Volume: The Dallas Heart Study. Circ Heart Fail. 2017 Aug;10(8):e003959. doi: 10.1161/CIRCHEARTFAILURE.117.003959. PMID 28775115
- [Derived] Cusano NE, Maalouf NM, Wang PY, Zhang C, Cremers SC, Haney EM, Bauer DC, Orwoll ES, Bilezikian JP. Normocalcemic hyperparathyroidism and hypoparathyroidism in two community-based nonreferral populations. J Clin Endocrinol Metab. 2013 Jul;98(7):2734-41. doi: 10.1210/jc.2013-1300. Epub 2013 May 20. PMID 23690312